CLINICAL TRIAL: NCT02024061
Title: Tratamento da Obesidade Pedi ́Atrica (TOP) - Uma Abordagem Multidisciplinar Envolvendo Pais e Pares
Brief Title: Treatment of Pediatric Obesity (TOP) - A Multidisciplinary Approach Involving Adolescents and Their Peers
Acronym: TOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Lusófona (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); University of Lisbon (Other)
Responsible Party: Principal Investigator, Antonio Palmeira, Associate Professor, Grupo Lusófona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTDC/DES/113591/2009
Record Dates: First submitted 2013-12-12; First posted 2013-12-31 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Obesity; Physical Activity; Sedentary Lifestyle
Keywords: Adolescents; Obesity; Physical activity; Sedentary behavior; Psychosocial health
MeSH Terms: conditions — Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer support (Experimental): The intervention will be similar with the exception that in the experimental group during the interventions (Interactive Sessions, Physical activity sessions and holiday camps), the presence of peers is predominant, indispensable and motivational in the context and the dynamics of development of activities.
  A team composed by a paediatrician and five exercise physiologists will conduct the delivery of the intervention. They all have previous training in adolescent obesity, resulting from their involvement in the adolescent obesity consult at the Hospital of Santa Maria.
  Interventions: Behavioral: Peer support
- Regular treatment (Active Comparator): The intervention will be similar with the exception that in the experimental group during the interventions (IS, PA sessions and holiday camps), the presence of peers is predominant, indispensible and motivational in the context and the dynamics of development of activities.
  A team composed by a paediatrician and five exercise physiologists will conduct the delivery of the intervention. They all have previous training in adolescent obesity, resulting from their involvement in the adolescent obesity consult at the Hospital of Santa Maria.
  Interventions: Behavioral: Regular treatment

INTERVENTIONS:
Behavioral: Peer support
  Arms: Peer support
Behavioral: Regular treatment — The participants in this arm will receive the regular obesity treatment provided by the hospital and university (interactive sessions and physical activity).
  Arms: Regular treatment

SUMMARY:
The purpose of this study is to analyse if a multidisciplinary approach including peers is effective in the treatment of obesity in adolescence.

DETAILED DESCRIPTION:
One in every 3 Portuguese adolescents is overweight (14% obese) (ONOCOP, 2009). Several institutions state that prevention is of upmost importance to deal with this epidemic (Council on Sports Medicine and Fitness; Council on School Health, 2006, August et al, 2008, Kohn et al, 2006), but public health stakeholders should also increase their efforts to treat those who already have excessive weight (Oude Luttikhuis et al, 2009). Several facts support this need, namely that obesity in adolescence: a) has a significant impact on both physical and psychosocial health (Lobstein et al, 2004); b) is an independent risk factor for adult obesity (Singh et al, 2008); c) is an independent risk factor for all cause mortality in adulthood - a more powerful predictor than being overweight in adult (Must et al, 1992); and d) is a major threat to the steady rise in life expectancy that occurred during the past two centuries (Olshansky et al, 2005).

Albeit this cumulative knowledge, treatment options remain elusive. A Cochrane review (Oude Luttikhuis et al, 2009) concluded that combined behavioral lifestyle interventions, when compared to standard care or self-help, provide significant and clinically meaningful reductions on weight in adolescents; and that the interventions should consider psychosocial determinants for behavior change and strategies to improve clinician-family interaction, in order to improve the desired outcomes.

The team of the TOP project has been working in this subject since 2004: the consult for obese adolescents of the Hospital de Santa Maria (HSM), a result of the collaboration between the two proponent Institutions. This has allowed the inclusion of exercise specialists in the obese adolescent' consult of the HSM, leading to an unusual (Fonseca et al, 2008), but surely necessary (Barlow et al, 2007), multidisciplinary program where, in the same Unit, adolescents are evaluated and receive medical, dietary and physical activity counselling. In compliance with the latest recommendations (Oude Luttikhuis et al, 2009), we use behavior change techniques directed not only to the adolescent but also to their parents, using the self-determination theory (SDT) rationale and motivational interviewing techniques (Teixeira et al, 2012), a treatment protocol that has been recognized by the Society for Adolescent Medicine (Fonseca et al, 2010).

Based on our previous experience and on recent literature that claims for the inclusion of peers as co-adjuvant on the weight management tasks, we hypothesize that: a) a larger and more frequent contact with the treatment staff; and b) the inclusion of peers as co-adjuvant on the weight management tasks in the TOP is necessary. Indeed, literature shows that adolescent' health related behaviors are associated with peer behaviors, in what Dishion named Social Contagion (Dishion & Dodge, 2005). Additionally, we think that regular physical activity (PA) and interactive educative sessions can provide the background to promote these two factors (Fonseca et al, 2012).

Therefore, the primary objective of this project is to develop, implement, and evaluate a treatment for adolescent obesity, which will use PA and interactive sessions to promote weight management skills, through the increase of contact time between the adolescent, parents, peers and treatment staff.

The primary outcomes will be body composition related variables, PA and sedentary behaviors. We will also look for putative moderators and mediators, derived from the behavior change rationales followed in the project, which will help understand and predict how the program has influenced the outcomes.

This project holds unique characteristics which comply with the latest recommendations for the treatment of adolescent obesity, and others that we have not been able to find in the literature: a) the inclusion of peers explicitly on the treatment protocol; b) the clinical setting of the treatment, with "real-life" subjects; c) objective measurements of the outcomes; d) the long-term treatment; and e) a well established rational (SDT and experiential learning) for the behavior change and to analyze the causal relations between predictors and outcomes.

This research is expected to contribute with increased knowledge about treatment options for adolescent obesity, specifically about the potential role of the inclusion of peers and increased time of contact through PA and interactive sessions. We also expect to contribute in a significant and clinically meaningful way to the weight management of the intervened adolescents. And, as HSM is a central hospital and a part of a medical university, the accumulated knowledge of the project will certainly be efficiently widespread to several other hospitals and obesity centers.

ELIGIBILITY:
Inclusion Criteria:

* Obese adolescents with BMI greater than or equal to the 95th percentile
* Aged between 14 and 17
* Caucasian
* Agree to the commitment.

Exclusion Criteria:

* Adolescents with serious illnesses
* Other factors preventing the engagement in regular PA

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in BMI z-score | Baseline, 4, 8 and 12 mo
  BMI z-score will be calculated through height and weight measured with standardised procedures
Change in % Fat Mass | Baseline, 6 and 12 mo
  The % of Fat Mass will be measured through dual energy x-ray absorptiometry.
Change in the Physical Activity Level | Baseline, 4, 8 and 12 mo
  The Physical Activity Level will be assessed by actigraphy (Actigraph GT3x).
Change in Sedentary behavior | Baseline, 4, 8 and 12 mo
  The sedentary behavior will be assessed by actigraphy (Actigraph GT3x) and by questionnaires (ASAQ)

SECONDARY OUTCOMES:
Changes in psychosocial health | Baseline, 4, 8 and 12 mo
  Quality of life, well-being and self-regulation variables will be measured by validated psychometric questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Helena R Fonseca, MD, PhD, Principal Investigator — Faculty of Medicine, University of Lisbon; Antonio L Palmeira, PhD, Principal Investigator — U. Lusófona Humanidades e Tecnologias
Locations (2):
- Portugal (2):
  - Consulta de Obesidade na Adolescência, Hospital Santa Maria, Lisbon
  - Universidade Lusófona Humanidades e Tecnologias, Lisbon

REFERENCES:
- [Background] ONOCOP, Study of the Pediatric and Adolescent Obesity Prevalence in Mainland Portugal - EPOBI. 2009, National Observatory of Obesity and Weight Control: Vilamoura - Portugal.
- [Background] Council on Sports Medicine and Fitness; Council on School Health. Active healthy living: prevention of childhood obesity through increased physical activity. Pediatrics. 2006 May;117(5):1834-42. doi: 10.1542/peds.2006-0472. PMID 16651347
- [Background] August GP, Caprio S, Fennoy I, Freemark M, Kaufman FR, Lustig RH, Silverstein JH, Speiser PW, Styne DM, Montori VM; Endocrine Society. Prevention and treatment of pediatric obesity: an endocrine society clinical practice guideline based on expert opinion. J Clin Endocrinol Metab. 2008 Dec;93(12):4576-99. doi: 10.1210/jc.2007-2458. Epub 2008 Sep 9. PMID 18782869
- [Background] Kohn M, Rees JM, Brill S, Fonseca H, Jacobson M, Katzman DK, Loghmani ES, Neumark-Sztainer D, Schneider M. Preventing and treating adolescent obesity: a position paper of the Society for Adolescent Medicine. J Adolesc Health. 2006 Jun;38(6):784-7. doi: 10.1016/j.jadohealth.2006.03.001. No abstract available. PMID 16761338
- [Background] Oude Luttikhuis H, Baur L, Jansen H, Shrewsbury VA, O'Malley C, Stolk RP, Summerbell CD. Interventions for treating obesity in children. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD001872. doi: 10.1002/14651858.CD001872.pub2. PMID 19160202
- [Background] Lobstein T, Baur L, Uauy R; IASO International Obesity TaskForce. Obesity in children and young people: a crisis in public health. Obes Rev. 2004 May;5 Suppl 1:4-104. doi: 10.1111/j.1467-789X.2004.00133.x. No abstract available. PMID 15096099
- [Background] Singh AS, Mulder C, Twisk JW, van Mechelen W, Chinapaw MJ. Tracking of childhood overweight into adulthood: a systematic review of the literature. Obes Rev. 2008 Sep;9(5):474-88. doi: 10.1111/j.1467-789X.2008.00475.x. Epub 2008 Mar 5. PMID 18331423
- [Background] Must A, Jacques PF, Dallal GE, Bajema CJ, Dietz WH. Long-term morbidity and mortality of overweight adolescents. A follow-up of the Harvard Growth Study of 1922 to 1935. N Engl J Med. 1992 Nov 5;327(19):1350-5. doi: 10.1056/NEJM199211053271904. PMID 1406836
- [Background] Olshansky SJ, Passaro DJ, Hershow RC, Layden J, Carnes BA, Brody J, Hayflick L, Butler RN, Allison DB, Ludwig DS. A potential decline in life expectancy in the United States in the 21st century. N Engl J Med. 2005 Mar 17;352(11):1138-45. doi: 10.1056/NEJMsr043743. PMID 15784668
- [Background] Fonseca H, Palmeira AL,Martins SS. Adolescent obesity: what we know and what we do. in Society for Adolescent Medicine Annual Meeting. 2008. Greensboro, EUA.
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Teixeira PJ, Silva MN, Mata J, Palmeira AL, Markland D. Motivation, self-determination, and long-term weight control. Int J Behav Nutr Phys Act. 2012 Mar 2;9:22. doi: 10.1186/1479-5868-9-22. PMID 22385818
- [Background] Fonseca H, Martins SS, Palmeira, AL. Institute: Assessment and treatment of overweight adolescents based on self-determination theory: A multidisciplinary program. in Society for Adolescent Medicine - 2010 Annual Meeting. 2010. Toronto - Canada.
- [Background] Dishion TJ, Dodge KA. Peer contagion in interventions for children and adolescents: moving towards an understanding of the ecology and dynamics of change. J Abnorm Child Psychol. 2005 Jun;33(3):395-400. doi: 10.1007/s10802-005-3579-z. PMID 15957566
- [Background] Fonseca H, Palmeira AL, Martins S, Ferreira PD. Short- and medium-term impact of a residential weight-loss camp for overweight adolescents. Int J Adolesc Med Health. 2014;26(1):33-8. doi: 10.1515/ijamh-2012-0107. PMID 23241665
- [Derived] Ascenso A, Palmeira A, Pedro LM, Martins S, Fonseca H. Physical activity and cardiorespiratory fitness, but not sedentary behavior, are associated with carotid intima-media thickness in obese adolescents. Eur J Pediatr. 2016 Mar;175(3):391-8. doi: 10.1007/s00431-015-2654-x. Epub 2015 Oct 21. PMID 26490566
- [Derived] Fonseca H, Palmeira AL, Martins SC, Falcato L, Quaresma A. Managing paediatric obesity: a multidisciplinary intervention including peers in the therapeutic process. BMC Pediatr. 2014 Apr 3;14:89. doi: 10.1186/1471-2431-14-89. PMID 24693926
- See also: Website that was used for the recruitment, currently under development to include the results and publications of the study — http://top.ulusofona.pt